CLINICAL TRIAL: NCT01651728
Title: Effect of Simvastatin on Pneumonia Prognosis in Elderly Patients: A Study of Immunological, Inflammatory, and Coagulation Responses in Relation to Reduce Mortality During Hospitalization
Brief Title: Effect of Simvastatin on Pneumonia Prognosis in Elderly Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Kuntjoro Harimurti, M.D., M.Sc., Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 48/PT02.FK/ETIK/2012; U1111-1133-2403 (Registry Identifier: International Clinical Trials Registry Platform (WHO-ICTRP))
Record Dates: First submitted 2012-07-24; First posted 2012-07-27 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Community-Acquired Pneumonia
Keywords: Simvastatin; Pneumonia; Elderly; TNF-α; IFN-ϒ; PAI-1; CRP
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simvastatin (Experimental): Tablet 20 mg once daily for 30 days
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): Placebo tablet once daily for 30 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — Tablet 20 mg once daily for 30 days
  Other Names: CAS Number 79902-63-9; ATC Code C10AA01
  Arms: Simvastatin
Drug: Placebo — daily for 30 days
  Arms: Placebo

SUMMARY:
The objective is to assess the effect of simvastatin on immunology, inflammatory, and coagulation responses, and mortality in elderly with pneumonia based. The primary outcome is mortality event.

The hypothesis of this study is that simvastatin therapy will reduce mortality in elderly with pneumonia.

DETAILED DESCRIPTION:
Elderly patients diagnosed with pneumonia after getting information and signing informed consent will be included in this trial. Simvastatin 20 mg will be administered to intervention group, while control group will receive placebo. Both groups will receive drugs (or placebo) for 30 days.

Baseline data will be collected within 24 hours after admission. Then the subject will be followed up for 30 days. At the 7th day, patients will be underwent several laboratory tests, i.e. serum TNF-α (Tumor Necrosis Factor alpha), IFN-ϒ Interferon gamma), CRP (C-Reactive Protein), and PAI-1 (Plasminogen Activator Inhibitor-1). Death from all causes until 30 days will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients with pneumonia

Exclusion Criteria:

* Severe septic condition
* Hepatic Cirrhosis
* Acute coronary disease
* Total cholesterol which is too high or too low
* In anticoagulant therapy
* In steroid therapy or other immunosuppressant therapy
* Have refused to join the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-08 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Death | 30 days

SECONDARY OUTCOMES:
Change from baseline in TNF-α (Tumor Necrosis Factor alpha) concentration | Baseline and 7 days
Change from baseline in Interferon-gamma (INF-ϒ) concentration | Baseline and 7 days
Change from baseline in Plasminogen Activator Inhibitor-1 (PAI-1) concentration | Baseline and 7 days
Change from baseline in C-Reactive Protein (CRP) concentration | Baseline and 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Kuntjoro Harimurti, MD, MSc, Principal Investigator — Department of Internal Medicine, Cipto Mangunkusumo Hospital, Faculty of Medicine University of Indonesia
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

REFERENCES:
- [Background] Dublin S, Jackson ML, Nelson JC, Weiss NS, Larson EB, Jackson LA. Statin use and risk of community acquired pneumonia in older people: population based case-control study. BMJ. 2009 Jun 16;338:b2137. doi: 10.1136/bmj.b2137. PMID 19531550
- [Background] Thomsen RW, Riis A, Kornum JB, Christensen S, Johnsen SP, Sorensen HT. Preadmission use of statins and outcomes after hospitalization with pneumonia: population-based cohort study of 29,900 patients. Arch Intern Med. 2008 Oct 27;168(19):2081-7. doi: 10.1001/archinte.168.19.2081. PMID 18955636